CLINICAL TRIAL: NCT07337044
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics in Healthy Adult Subjects After Subcutaneous Injection of TISA-818-Inj
Brief Title: Evaluate the Safety, Tolerability, and Pharmacokinetics in Healthy Adult Subjects After Subcutaneous Injection of TISA-818-Inj
Acronym: TISA-818-Inj
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EnliTISA (Shanghai) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TISA-818-22101
Record Dates: First submitted 2025-12-07; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects
Keywords: Phase 1 clinical study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TISA-818-Inj group (Experimental)
  Interventions: Drug: TISA-818-Inj
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TISA-818-Inj — TISA-818-Inj
  Arms: TISA-818-Inj group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This is a single-centre, randomised, double-blind, placebo-controlled, dose escalation study to assess the safety, tolerability, and pharmacokinetic (PK) profile, of TISA-818-Inj-5mg/mL after single and multiple s.c. injections in healthy subjects.

The study consisted of two parts： Part A: Single ascending dose (SAD) in healthy adult subjects (3 dose cohorts, 6 active and 2 placebo/cohort) Part B: Multiple ascending dose (MAD) with 7 days once daily administration in healthy adult subjects (3 dose cohorts, 6 active and 2 placebo/cohort)

ELIGIBILITY:
Inclusion criteria

1. Willing and able to give written informed consent for participation in the study.
2. The subject is considered by the Investigator to be in good general health as determined by medical history, clinical laboratory test results, vital signs measurements, 12-lead ECG results, and physical examination findings at screening.
3. For all women of childbearing potential (WOCBP) a negative pregnancy test at screening and a negative urine dip-stick pregnancy test at baseline, prior to first dose of Investigational medicinal product (IMP) will be required.
4. Females of non-childbearing potential must have documented tubal ligation or hysterectomy; or be post-menopausal (defined as 12 months of amenorrhoea [in questionable cases a blood sample with follicle stimulating hormone (FSH) 25-140 IE/L is confirmatory]).
5. WOCBP must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy from at least 4 weeks prior to dose until 30 days after (last) IMP administration. Their male partner must agree to use a condom during the same time frame.
6. Fertile male subjects must be willing to use condom and assure that their fertile female partner will use contraceptive methods with a failure rate of < 1% 12 to prevent pregnancy and drug exposure of a fertile female partner and refrain from donating sperm from the date of dosing until 30 days after dosing of the IMP. Men who are surgically sterile may be included without they/their partner fulfilling the above criteria on birth control.

Exclusion criteria

1. Current evidence or history of clinically significant (as judged by the Investigator) haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including asthma, chronic obstructive pulmonary disease [COPD] and drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
3. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the study.
5. History of severe allergy/hypersensitivity or on-going allergy/hypersensitivity (such as seasonal allergy, pet allergy, allergy to a different class of drug etc.), as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to TISA-818.
6. History of severe COVID-19 infection requiring hospitalisation within the last 12 months prior to screening, or clinical history compatible with Long COVID-19 (symptoms beyond 12 weeks of acute infection).
7. Administration of a live viral vaccine (e.g. measles-mumps-rubella, varicella zoster, herpes zoster, oral polio virus, FluMist, attenuated typhoid fever vaccine, or attenuated rotavirus vaccine) within 8 weeks prior to screening and/or is unwilling to avoid live viral vaccines for at-least 8 weeks following completion of the final study visit.
8. Prolonged QTcF (>450 ms for men, >470 ms for women), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
9. After 10 min supine rest at the time of screening, any vital signs values outside the following ranges:

   1. Systolic blood pressure < 90 mmHg or ≥ 140 mmHg, or
   2. Diastolic blood pressure < 50 mmHg or ≥ 90 mmHg, or
   3. Pulse <40 or >90 beats per min (bpm)
10. Any positive result on screening for human immunodeficiency virus (HIV), hepatitis B (serum hepatitis B surface antigen positive), hepatitis C (e.g. HCV RNA positive).
11. Any clinically significant abnormal safety laboratory values, as judged by the Investigator.
12. Current smoker or user of nicotine products. Irregular use of nicotine (e.g. smoking, snuffing, chewing tobacco) less than three times per week is allowed before Day -1.
13. Positive screening result for drugs of abuse or alcohol at the time of screening or on admission to the clinic prior to administration of the IMP.
14. Subjects who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the study.
15. History of binge drinking or frequent alcohol consumption within 6 months prior to the study (more than 14 units of alcohol per week, 1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine).
16. Any present or historic use of drugs of abuse or anabolic steroids.
17. Frequent excessive consumption of tea, coffee, or caffeinated beverages (more than 5 cups a day, 1 cup = 200 ml) in the 3 months prior to screening or ingestion of any food or drink containing caffeine , alcohol, xanthine, or grapefruit within 48 hours prior to randomisation.
18. Inability to be venepunctured and/or tolerate venous access.
19. Inability or un-willingness to be administered the number of s.c. injections to be given in applicable dose cohort (e.g. afraid of needled/sticks, unhealthy skin, or too skinny), as judged by the Investigator.
20. Blood donation (or corresponding blood loss) ≥ 450 mL of blood within 3 months before Day -1 (except for female menstrual blood loss), or plan to donate blood or blood components during the study or within 3 months after the end of the study.
21. Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins, and minerals within 2 weeks prior to (first) administration of IMP. Use of montelukast sodium and other leukotriene receptor inhibitors is not allowed during the same period.
22. Any medications or herbal remedies, including St John's Wort, known to chronically alter drug absorption or elimination processes within 4 weeks prior to first IMP administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
23. Administration of another new chemical entity (defined as a compound that has not been approved for marketing) or has participated in any other clinical study that included drug treatment with the last administration within 3 months prior to administration of IMP in this study. Subjects consented and screened but not dosed in previous phase 1 studies are not excluded.
24. Investigator considers the subject unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Frequency, intensity, and seriousness of Treatment Emergent Adverse Events | UP to 20 days
  Frequency, intensity, and seriousness of adverse events following subcutaneous injection of TISA-818.

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters of TISA-818 following a single-dose and multiple-doses of TISA-818 injection | Up to 72 hours
  For PK analysis, blood samples will be collected before and up to 72 hours after the subcutaneous injection of TISA-818 to determine TISA-818 serum concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
The result of this trial will not be published in the International Committee of Medical Journal.